CLINICAL TRIAL: NCT05711069
Title: The Effect of Core Stabilization Exercise Program on Kicking Velocity, Sprint Speed and Agility Performance in Male Adolescent Football Players
Brief Title: Core Stabilization Programme on Kicking Velocity and Performance in Male Adolescent Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyda Sofuoğlu, Principal investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETK00-2020-0243
Record Dates: First submitted 2022-10-22; First posted 2023-02-02 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Soccer; Core Stability; Sports Performance
Keywords: Exercise; Core Stability; Kicking velocity; Run Speed; Agility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Exercise Program Group (Active Comparator): 23 Football players from Gönyeli Futbol Akademisi voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. Athletes will involve 8 Weeks core stability exercise program. During this process they will continue to attend routine football training program. After 8. Weeks assessments will be repeated.
  Interventions: Other: Core Stability Exercise Program
- Routine Football Training Program Group (Other): 22 Football players from Gönyeli Futbol Akademisi voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. Kicking velocity, run speed and agility performance will evaluate and athletes will continue to attend football training program. After 8 Weeks assessments will be repeated.
  Interventions: Other: Routine Football Training Program

INTERVENTIONS:
Other: Core Stability Exercise Program — Core stability is an important component maximising efficient athletic function. Function is most often produced by the kinetic chain, the coordinate sequenced activation of body segments that places the distal segment in the optimum position at the optimum velocity with the optimum timing to produce the desired athletic task. Speed and power are critical performance factors in football. Football including jumping, kicking, tackling, turning, sprinting, changing pace, and sustaining forceful contractions to maintain balance and control of the ball against defensive pressure. İn the literature, no study has demonstrated the effectiveness of core stability exercise program in adolescent football players.
  Arms: Core Stability Exercise Program Group
Other: Routine Football Training Program — Core stability is an important component maximising efficient athletic function. Function is most often produced by the kinetic chain, the coordinate sequenced activation of body segments that places the distal segment in the optimum position at the optimum velocity with the optimum timing to produce the desired athletic task. Speed and power are critical performance factors in football. Football including jumping, kicking, tackling, turning, sprinting, changing pace, and sustaining forceful contractions to maintain balance and control of the ball against defensive pressure. İn the literature, no study has demonstrated the effectiveness of core stability exercise program in adolescent football players.
  Arms: Routine Football Training Program Group

SUMMARY:
Core stability is an important component maximising efficient athletic function. Function is most often produced by the kinetic chain, the coordinate sequenced activation of body segments that places the distal segment in the optimum position at the optimum velocity with the optimum timing to produce the desired athletic task. Speed and power are critical performance factors in football. Football including jumping, kicking, tackling, turning, sprinting, changing pace, and sustaining forceful contractions to maintain balance and control of the ball against defensive pressure. In the literature, no study has demonstrated the effectiveness of core stability exercise program in adolescent football players.The aim of this study was to evaluate the effectiveness of core stabilization exercise program on adolescent male football players.

DETAILED DESCRIPTION:
Core stability is an important component maximising efficient athletic function. Function is most often produced by the kinetic chain, the coordinate sequenced activation of body segments that places the distal segment in the optimum position at the optimum velocity with the optimum timing to produce the desired athletic task. The importance of core stability for injury prevention and performance enhancement has been popularized during the past decades. Up to date, core muscle strengthening plays an important role in different prevention programs, such as the "FIFA 11 +". Football is considered a high-intensity intermittent sport requiring high levels of physical fitness related to the ability to perform powerful actions, with a varied range of activities that involve both breaking and propulsive forces as well as distinct contraction modes and velocities. Speed and power are critical performance factors in football. Football including jumping, kicking, tackling, turning, sprinting, changing pace, and sustaining forceful contractions to maintain balance and control of the ball against defensive pressure. Kicking is one of the most fundamental and frequently used skills in soccer and its motion consists of several stages as follows: (1) the withdrawal of the thigh and shank (backswing); (2) the forward rotation of the thigh and shank, which occurs as a result of hip flexion; (3) the reduction of thigh angular velocity, with a corresponding increase in shank angular velocity up to impact with the ball; and (4) the follow-through. Football is seen as highly intensive sport with an increased injury rate. In adolescent football players, muscle-tendon unit adaptation is effecting by athletic performance. The mechanic loading on this unit results increase risk of lower extremity injuries. In the literature, no study has demonstrated the effectiveness of core stability exercise program in adolescent football players.The aim of this study was to evaluate the effectiveness of core stabilization exercise program on adolescent male football players.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are not get any operation related with lower extremity and spine in last 6 months.
* Subjects who are voluntary to participate in the study and get informed consent form from legal representative.
* Subjects who attend in football training regularly.

Exclusion Criteria:

* Current pain in lower extremity and spine.
* Subjects who have discontinuity in training program or exercise program more than 3 times.
* Subjects who have difficulty to apply exercise program.

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volga Bayrakcı Tunay, Prof, Study Director — Hacettepe University
Locations (1):
- Fizyo osteopati Fizik Tedavi ve Sağlıklı Yaşam Merkezi, Nicosia, Lefkoşa, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
IPD data for all primary and secondary measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 1 year of study publication.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Stability Exercise Program Group: 23 Football players from Gönyeli Futbol Akademisi voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. Before implementing the core stability exercise program, participants' ball-kicking velocity, sprint speed, and agility performance will measure with a Bushnell velocity radar gun, 20 m sprint test, and 505 agility test. Athletes will involve 8 Weeks core stability exercise program. During this process they will continue to attend routine football training program. After 8 Weeks core stability exercise program assessments will be repeated.
  Core Stability Exercise Program: Core stability is an important component maximising efficient athletic function. Function is most often produced by the kinetic chain, the coordinate sequenced activation of body segments that places the distal segment in the optimum position at the optimum velocity with the optimum timing to produce the desired athletic task. Speed and power are critical performance factors in football. Football including jumping, kicking, tackling, turning, sprinting, changing pace, and sustaining forceful contractions to maintain balance and control of the ball against defensive pressure. İn the literature, no study has demonstrated the effectiveness of core stability exercise program in adolescent football players.
- Routine Football Training Program Group: 22 Football players from Gönyeli Futbol Akademisi voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. Ball-kicking velocity, sprint speed, and agility performance will measure with a Bushnell velocity radar gun, 20 m sprint test, and 505 agility test. Athletes will continue to attend only routine football training program. After 8 Weeks assessments will be repeated.
  Routine Football Training Program: This group will continue to routine football training program with their coach 3 times a week.
Period: Overall Study
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group
Started | 23 | 22
Completed | 19 | 17
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 17 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 17 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Cyprus | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Kicking Velocity Measurement
Description: Kicking velocity will measure with Bushnell Velocity Radar Gun ((Bushnell Performance Optics, Overland Park, KS) in km/h.
Time Frame: Measurement will repeat three times in 2 minutes intervals and the mean value will be taken. Baseline and 8 Weeks reported.
Population: 4 participants from core stability exercise program group and 5 participants from routine football training program group were excluded from the study due to did not fullfilled inclusion criteria. 19 participants from core stability exercise prpgram group and 17participants from routine football training program group were included to the study.
Measure: Mean (Standard Deviation); unit: KM/H
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group
Number analyzed (Participants) | 19 | 17
KM/H
  Baseline | 71.89 (16.21) | 67.71 (13.80)
  8 Weeks | 81.05 (8.46) | 69.12 (13.04)

2. Primary Outcome: Run Speed Measurement
Description: Run speed will measure with 20 Meter Sprint Test in sec.
Time Frame: Measurement will repeat three times in 2 minutes intervals and mean value will be taken. Baseline and 8 Weeks reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group
Number analyzed (Participants) | 19 | 17
Second
  Baseline | 3.86 (0.40) | 3.96 (0.25)
  8 Weeks | 3.60 (0.23) | 3.95 (0.34)

3. Primary Outcome: Agility Measurement
Description: Agility will measure with 505 Agility Test in sec. The athlete runs from the 15 meter marker towards the line and through the 5 m markers, turns on the line and runs back through the 5 meter marker and stopped when they return through these markers (that is, the time taken to cover the 5 m up and back distance -10 m total).
Time Frame: Measurements will repeat three times in 2 minutes intervals and mean value will be taken. Baseline and 8 Weeks reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group
Number analyzed (Participants) | 19 | 17
Second
  Baseline | 3.03 (0.28) | 3.03 (0.20)
  8 Weeks | 2.80 (0.28) | 2.93 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 10 weeks.
Arm/Group | Core Stability Exercise Program Group | Routine Football Training Program Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 4/23 | 5/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Stability Exercise Program Group (N=23) | Routine Football Training Program Group (N=22)
Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Discontinuity (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT05711069/Prot_SAP_000.pdf